CLINICAL TRIAL: NCT03906864
Title: Integrated Care Pathway for Hip Fractures in a Subacute Rehabilitation Setting
Brief Title: Care Pathway for Sub-acute Hip Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Luke's Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Boon Yeow, Tan, Chief Executive Officer, Medical Director, Medical Division, St Luke's Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: slhdoc01; 65 68953250 (Other: St Luke's Hospital)
Record Dates: First submitted 2018-09-16; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hip Fractures
Keywords: Critical pathway, length of stay, recovery of function, subacute care
MeSH Terms: conditions — Hip Fractures | interventions — Critical Pathways

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual care consisted of 2 half hourly therapy sessions per day from Monday to Friday and medical ward rounds 3 times a week. Multidisciplinary rounds were conducted every 2 weeks. Any specific goals or interventions were at the discretion of the managing team.
- Intervention group (Experimental): Intervention group had structured assessments and checklists (as part of the integrated care pathway) in addition to usual care.
  Interventions: Other: Care Pathway

INTERVENTIONS:
Other: Care Pathway — The intervention group had the following as part of the integrated care pathway:
  1. Medical assessment on admission for risk factors for falls.
  2. A weekly assessment of complications including pain, deep venous thrombosis, anaemia, wounds and pressure ulcers, etc. The Confusion Assessment Method and the Geriatric Depression Scale were utilized.
  3. Physiotherapy and occupational therapy guidelines with recommended milestones (set for the full, partial and non-weight bearing groups)
  4. Physiotherapy Clinical Outcome Variables Scale (PTCOVS)16 was used by the physiotherapists in the intervention group to assess the baseline mobility, to define outcome goals and to direct treatment plans.
  5. A postoperative hip precaution handout (containing information on avoiding hip prosthesis dislocation in patients with total hip replacement or hemiarthroplasty) was given to patients and their caregivers.
  Arms: Intervention group

SUMMARY:
The effectiveness of integrated care pathways for hip fractures in sub-acute rehabilitation settings is not known. The study objective was to assess if a hip fracture integrated care pathway at a sub-acute rehabilitation facility would result in better functional outcomes, shorter length of stay and fewer institutionalisations. A randomised controlled trial on an integrated care pathway was conducted for hip fracture patients in a sub-acute rehabilitation setting. The study supports the use of integrated care pathways in sub-acute rehabilitation settings to reduce length of stay whilst achieving the same functional gains.

DETAILED DESCRIPTION:
All patients admitted to St Luke's Hospital, a 185-bed hospital in Singapore providing multidisciplinary stepdown care, from 8 September 2004 to 14 June 2006 for the purpose of rehabilitation after a new hip fracture were included. Patients were excluded if any of the following criteria were present: (i) Pre-morbid non-ambulatory status, (ii) nursing home residents, (iii) palliative care patients, and (iv) patients previously enlisted for the trial. Administrative staff allocated patients to either ICP or usual care according to the last digit of their National Registration Identity Card (NRIC) numbers, odd numbers to the intervention group and even numbers to the control group. Patients were then admitted to 1 of 2 intervention wards or 1 of 3 control wards. Patients were enrolled by the principal investigators only after moving into their respective wards because of work flow limitations. Those who refused consent or were excluded remained in their assigned wards and received usual care. Both intervention and control groups were under the care of multidisciplinary teams but the intervention group had structured assessments and checklists in addition to usual care while the control group had usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to St Luke's Hospital for the purpose of rehabilitation after a new hip fracture.

Exclusion Criteria:

* Patients were excluded if any of the following criteria were present: (i) Pre-morbid non-ambulatory status, (ii) nursing home residents, (iii) palliative care patients, and (iv) patients previously enlisted for the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2004-09-08 (Actual); Primary Completion 2006-06-14 (Actual); Study Completion 2012-12-26 (Actual)

PRIMARY OUTCOMES:
Montebello Rehabilitation Factor Score (MRFS) | 1 day At discharge
  MRFS is a recognised measure of hip fracture patients' functional outcome, calculated with the following formula, using the Modified Barthel Index (MBI) scores (which scores the degree of independence of a subject from any assistance up to a maximum score of 100)
Montebello Rehabilitation Factor Score (MRFS) | At 6 months
  MRFS is a recognised measure of hip fracture patients' functional outcome, calculated with the following formula, using the Modified Barthel Index (MBI) scores (which scores the degree of independence of a subject from any assistance up to a maximum score of 100)
Montebello Rehabilitation Factor Score (MRFS) | At 1 year
  MRFS is a recognised measure of hip fracture patients' functional outcome, calculated with the following formula, using the Modified Barthel Index (MBI) scores (which scores the degree of independence of a subject from any assistance up to a maximum score of 100)
Proportions of patients achieving pre-morbid ambulatory status | 1 day At discharge
  Pre-morbid ambulatory status is a predictor for post-operative mobility
Proportions of patients achieving pre-morbid ambulatory status | At 6 months
  Pre-morbid ambulatory status is a predictor for post-operative mobility
Proportions of patients achieving pre-morbid ambulatory status | At 1 year
  Pre-morbid ambulatory status is a predictor for post-operative mobility
Length of stay in hospital | 1 day At discharge
  Refers to the average number of days that patients spend in hospital
Percentage of patients admitted to nursing home | Up to 1 year after discharge
  A form of institutional care

SECONDARY OUTCOMES:
Readmissions to an acute hospital for any reason | up to 1-year post-discharge
  An episode when a patient who had been discharged from a hospital is admitted again within a specified time interval
Cumulated mortality | 1 year
  Probability or risk of individuals dying from the disease during a specified period
Quality of life scale-Short form 12 quality of life | 6 months and 1 year
  Scale for short form 12 quality of life 0-100
  Scale for Physical Component Summary (PCS) and Scale for Mental Component Summary (MCS), a multipurpose, generic measure of health status 0-100
  Interpretation of the score : The higher score, the better

CONTACTS AND LOCATIONS:
Overall Officials: Tze Pin Ng, FAMS, PhD, Study Chair — National University of Singapore
Locations (1):
- St Luke's Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330